CLINICAL TRIAL: NCT05757570
Title: Open-Label Study to Assess the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Povetacicept in Subjects With Autoimmune Cytopenias (RUBY-4)
Brief Title: An Open-label Study of Povetacicept in Participants With Autoimmune Cytopenias
Acronym: RUBY-4
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AIS-D04; 2023-507067-19-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia; Idiopathic Thrombocytopenic Purpura; Warm Autoimmune Hemolytic Anemia; Cold Agglutinin Disease
Keywords: Immune Thrombocytopenia; Warm Autoimmune Hemolytic Anemia; Cold Agglutinin Disease; Autoimmune Cytopenia; Idiopathic Thrombocytopenic Purpura; Immune Thrombocytopenic Purpura; Hemolytic Anemia; RUBY4; RUBY-4; Povetacicept; ALPN-303; ALPN303; Autoimmune Hemolytic Anemia; ITP; wAIHA; AIHA; CAD
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Anemia, Hemolytic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Povetacicept 240mg (Experimental): Participants grouped in 3 cohorts by diagnosis will be administered Povetacicept
  Interventions: Drug: povetacicept
- Part 2: Povetacicept Dose A (Experimental): Based on the findings of Part 1, one or two dose levels may be assessed in Part 2; if two dose levels are assessed participants will be randomized to receive one of the two dose levels of Povetacicept
  Interventions: Drug: povetacicept

INTERVENTIONS:
Drug: povetacicept — Administered by subcutaneous injection every 4 weeks
  Other Names: ALPN-303

SUMMARY:
The goal of this clinical study is to evaluate povetacicept in adults with autoimmune cytopenias of immune thrombocytopenia, autoimmune hemolytic anemia, and cold agglutinin disease to determine if povetacicept is safe and potentially beneficial in treating these diseases. During the study treatment period participants will receive povetacicept approximately every 4 weeks for 6 months, with the possibility of participating in a 6-month study treatment extension period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Indication-specific Criteria

   1. Immune Thrombocytopenia (ITP)

      * Documented persistent or chronic primary ITP of at least 12 weeks duration from diagnosis to Cycle 1 Day 1
      * History of failure or relapse to at least 2 treatment regimens for ITP
      * History of exposure to a TPO-RA unless otherwise contraindicated or unavailable
      * Documented history of platelets <30 × 10^9/L
   2. Warm Autoimmune Hemolytic Anemia (wAIHA)

      * Diagnosis of primary wAIHA of at least 12 weeks duration documented with a current or prior positive direct antiglobulin test (DAT) for anti-IgG (±C3d)
      * Documented history of anemia with hemoglobin ≤10 g/dL
      * At least one of the following: (i) haptoglobin < lower limit of normal (LLN) (ii) indirect bilirubin > upper limit of normal (ULN) (iii) lactate dehydrogenase>ULN
      * History of failure or relapse to at least 2 treatment regimens for wAIHA
   3. Cold Agglutinin Disease (CAD)

      * Diagnosis of primary CAD of at least 12 weeks duration with all of the following: (i) chronic hemolysis (ii) polyspecific DAT positive (iii) monospecific DAT strongly positive for C3d (iv) cold agglutinin titer ≥64 at 4°C (v) IgG DAT ≤1+ (vi) no overt malignant disease
      * Documented history of anemia with hemoglobin ≤10 g/dL
      * Evidence of hemolysis during screening: (i) indirect bilirubin >ULN and (ii) lactate dehydrogenase>ULN or haptoglobin <LLN
      * History of failure or relapse to at least 1 treatment regimen for CAD
2. (All indications) If receiving protocol-specified standard-of-care medications, doses must be stable for protocol-specified durations

Key Exclusion Criteria:

1. Secondary AIHA, CAD, or ITP
2. Treatment with any of the following within the noted period prior to study entry

   1. rituximab: <12 weeks
   2. IVIg: <4 weeks
   3. sutimlimab, any use after initiation of screening is exclusionary
   4. plasmapheresis, plasma exchange, or double-filtration plasmapheresis: <8 weeks
   5. transfusions with blood, blood products or other rescue medications: <2 weeks
   6. splenectomy: <12 weeks
   7. other immunomodulatory or investigational agents, except for investigational agents for COVID-19 that have been granted emergency use authorization or approved by the applicable national health authority: <5 half-lives and requires agreement of the Medical Monitor
3. Recent serious or ongoing infection; risk or history of serious infection

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Adverse events (AEs) and Serious adverse events (SAEs) | Study Day 1 through 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Locations (44):
- United States (15):
  - Investigational Site (230), Los Angeles, California
  - Investigational Site (401), Washington D.C., District of Columbia
  - Investigational Site (419), Cooper City, Florida
  - Investigational Site (425), Miami, Florida
  - Investigational Site (219), Iowa City, Iowa
  - Investigational Site (435), Columbia, Maryland
  - Investigational site (405), Lake Success, New York
  - Investigational Site (423), New Hyde Park, New York
  - Investigational Site (421), New York, New York
  - Investigational Site (404), New York, New York
  - Investigational Site (420), Shirley, New York
  - Investigational Site (422), The Bronx, New York
  - Investigational Site (414), Charlotte, North Carolina
  - Investigational Site (402), Greenville, North Carolina
  - Investigational Site (411), Seattle, Washington
- Australia (6):
  - Investigational Site (410), Box Hill
  - Investigational Site (519), Concord
  - Investigational Site (517), Douglas
  - Investigational Site (413), Liverpool
  - Investigational Site (407), West Perth
  - Investigational Site (409), Westmead
- Investigational Site (434), Vienna, Austria
- Canada (3):
  - Investigational Site (406), Greenfield Park
  - Investigational Site (403), Hamilton
  - Investigational Site (444), Toronto
- Investigational Site (438), Essen, Germany
- Italy (4):
  - Investigational Site (432), Meldola
  - Investigational Site (428), Milan
  - Investigational Site (431), Novara
  - Investigational Site (443), Trieste
- Norway (2):
  - Investigational Site (433), Grålum
  - Investigational Site (437), Trondheim
- Spain (5):
  - Investigational Site (436), Barcelona
  - Investigational Site (429), Burgos
  - Investigational Site (430), Madrid
  - Investigational Site (426), Murcia
  - Investigational Site (427), Seville
- Turkey (Türkiye) (3):
  - Investigational Site (415), Ankara
  - Investigational Site (416), Ankara
  - Investigational Site (418), Istanbul
- United Kingdom (4):
  - Investigational Site (442), Leeds
  - Investigational Site (439), London
  - Investigational Site (441), London
  - Investigational Site (440), London